CLINICAL TRIAL: NCT00853580
Title: A Randomized Placebo-Controlled Study of Lovastatin in Children With Neurofibromatosis Type 1
Acronym: STARS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Boston Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Children's National Research Institute (Other); Children's Hospital Medical Center, Cincinnati (Other); National Cancer Institute (NCI) (NIH); University of Chicago (Other); University of Utah (Other); Washington University School of Medicine (Other); Sydney Children's Hospitals Network (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Bruce Korf, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X080929007; DOD: W81XWH-05-1 0615 (Other: Department of Defense)
Record Dates: First submitted 2009-02-23; First posted 2009-03-02 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis Type 1, Neurocognitive, Phase II
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): This is a prospective multi-centre randomized, placebo-controlled Phase II study to determine the efficacy of Lovastatin ™ on visual spatial learning and/or attention abilities of children with NF1 aged between 8 and less than 16 years. In addition, the effect of Lovastatin ™ on secondary measures of executive function, visual spatial skills, behavior and quality of life will be assessed. Participants will be randomized to 16-weeks of treatment with Lovastatin ™ or a matched placebo.
  Interventions: Device: placebo
- 1 (Experimental): This is a prospective multi-centre randomized, placebo-controlled Phase II study to determine the efficacy of Lovastatin ™ on visual spatial learning and/or attention abilities of children with NF1 aged between 8 and less than 16 years. In addition, the effect of Lovastatin ™ on secondary measures of executive function, visual spatial skills, behavior and quality of life will be assessed. Participants will be randomized to 16-weeks of treatment with Lovastatin ™ or a matched placebo.
  Interventions: Drug: Lovastatin ™

INTERVENTIONS:
Drug: Lovastatin ™ — Lovastatin starting at 20mg for 2 weeks, increasing to 40mg for 14 weeks. Total duration of trial is 16 weeks.
  Arms: 1
Device: placebo — Starting at 20mg for 2 weeks, then increasing to 40mg for 14 additional weeks for a total duration of treatment of 16 weeks.
  Arms: 2

SUMMARY:
The specific aim of this study is to determine whether Lovastatin ™ significantly improves visual spatial learning and/or sustained attention in children with NF1.

Secondary Aims:

To evaluate the effect of Lovastatin ™ on measures of executive function, behavior and quality of life in children with NF1 and cognitive deficits.

To further evaluate the toxicity and tolerability of Lovastatin ™ in children with NF1 and cognitive deficits.

Hypotheses

It is hypothesized that Lovastatin ™ will improve the visual spatial memory and/or attention deficits in children with NF1. This is based on studies demonstrating that Lovastatin ™ has significantly improved impairments in visual spatial memory and attention in the NF1 murine model.

It is further expected that Lovastatin ™ will be safe and well tolerated over a 16-week period.

DETAILED DESCRIPTION:
Study Design

This is a prospective multi-centre randomized, placebo-controlled Phase II study to determine the efficacy of Lovastatin ™ on visual spatial learning and/or attention abilities of children with NF1 aged between 8 and less than 16 years. In addition, the effect of Lovastatin ™ on secondary measures of executive function, visual spatial skills, behavior and quality of life will be assessed. Participants will be randomized to 16-weeks of treatment with Lovastatin ™ or a matched placebo. It is plausible and ethical to employ a placebo group as no standard therapy with established efficacy is being withheld. There is no cross-over in this study due to a lack of data concerning the length of possible washout effects. The Lovastatin ™ dose will begin at 20 mg once daily/continuous dosing and escalate over a two-week period to 40 mg once daily/continuous dosing and continue at this dose for 14 weeks. Participants will be carefully monitored for side effects. The safety of Lovastatin ™ will be evaluated using laboratory tests, clinical signs and adverse effects, which will be monitored at regular intervals over the 16-week period. Primary and secondary outcome measures will be administered at baseline, 16 weeks post-treatment and at follow-up, 8 weeks after cessation of treatment to determine any carry-over effects. The safety of Lovastatin ™ will also be evaluated, with regular monitoring of side-effects during the trial.

Study Population

This is a Phase II study involving children with NF1 (aged between 8 years to 15 years 11 months old at time of enrollment) with evidence of cognitive impairment, defined as having a score of at least one standard deviation or more below the population mean on a measure of visual spatial learning and/or attention.

A total of 142 participants with NF1 aged between 8 years and 15 years 11 months will be enrolled in the study. The age limits were selected on the basis that Lovastatin ™ has been shown to be safe in children aged between 8 and 17 years old. In addition, one of the primary outcome measures (attention) only has normative data for up to 15 years 11 months. Therefore, the maximum age limit for participants at time of enrolment is 15 years 11 months so that normative data can be used to determine whether participants are impaired. The pediatric NF1 population is an ideal group in which to study the cognitive effects of Lovastatin ™ because it represents an opportunity for early pharmacological intervention of cognitive deficits.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged between 8 years and 15 years 11 months at time of enrollment who meet NIH diagnostic criteria for NF1 (Appendix 1)
* Participants must have a full-scale IQ of 70 or above. In cases where there is a statistically significant difference between verbal IQ and performance IQ (.05 level as determined by Table B3 in the WASI manual), participants will be eligible if at least one of these quotients is 70 or above
* Participants must have a cognitive impairment defined as having a score of at least one standard deviation or more below the population mean on one or more of the primary objective outcome measures (i.e., impaired on a measure of visual spatial learning and/or sustained attention)
* Participants must be medically stable
* Participants who are on a stable dose of methylphenidate and/or dextroamphetamines for at least one month prior to screening and who will remain on the same dose for the duration of the study.
* Hepatic function: Participants must have a bilirubin within normal limits and AST and ALT ± 2 times the upper limit of normal as determined by the standards at their institution
* Renal function: Participants must have an age-adjusted normal serum creatinine or a creatinine clearance of greater than 70 ml/m/1.73m2
* Hematologic function: Participants must have an absolute neutrophil count of greater than 1,500, a hemoglobin of greater than 9 gms/dl, and a platelet count of greater than 100,000 on study entry
* Participants must sign all required documents, including informed assent and HIPAA documents
* Female participants of childbearing age should not be pregnant, must have a negative pregnancy test before initiation of treatment, and take appropriate birth control precautions to participate in this study.

Exclusion Criteria:

* Full-scale IQ less than 70; In cases where this is a statistically significant difference between performance IQ and verbal IQ (.05 level), patients will be excluded if both quotients fall below 70
* Individuals that are not cognitively impaired on at least one of the primary objective outcome measures
* Individuals with insufficient English to complete the assessments
* Participants taking psychotropic medication other than methylphenidate and/or dextroamphetamines. These patients are eligible if, as clinically indicated, they cease medication for at least 30 days prior to screening and remain off these medication for the duration of the study
* Participants with intracranial pathology such as epilepsy, diagnosed head injury, hydrocephalus or progressive intracranial tumors (children with asymptomatic or static lesions will be eligible)
* Participants who are pregnant or breastfeeding; Participants who have received any investigational drug, other than sirolimus, within 30 days of initiation of study
* Participants who have recently taken Lovastatin. These participants will be eligible after a washout period of at least three months.
* Participants with significant hepatic, renal or hematologic function as previously defined
* Participants with a history of neuromuscular disease, excluding hypotonias thought to be associated with NF1
* Participants with a clinically significant unrelated illness, which in the judgment of the principal or associate investigator, would compromise the participant's ability to tolerate the medication or potentially interfere with the participant's ability to participate in the required testing
* Low cholesterol (lower limit of a total cholesterol of 90mg/dl)
* Participants who have recently taken sirolimus within three months of enrollment. These participants will be eligible after a washout period of at least three months.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2009-07; Primary Completion 2014-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn North, MD, Principal Investigator — University of Sydney - Westmead; Maria Acosta, MD, Study Director — Children's National Research Institute; Jonathan Payne, MD, Study Director — University of Sydney - Westmead
Locations (12):
- United States (11):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - NIH, Bethesda, Maryland
  - Children' Hospital Boston, Boston, Massachusetts
  - Washington University - St. Louis, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Medical Center - Univ. of Texas SW Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
- The Children's Hospital at Westmead, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Payne JM, Barton B, Ullrich NJ, Cantor A, Hearps SJ, Cutter G, Rosser T, Walsh KS, Gioia GA, Wolters PL, Tonsgard J, Schorry E, Viskochil D, Klesse L, Fisher M, Gutmann DH, Silva AJ, Hunter SJ, Rey-Casserly C, Cantor NL, Byars AW, Stavinoha PL, Ackerson JD, Armstrong CL, Isenberg J, O'Neil SH, Packer RJ, Korf B, Acosta MT, North KN; NF Clinical Trials Consortium. Randomized placebo-controlled study of lovastatin in children with neurofibromatosis type 1. Neurology. 2016 Dec 13;87(24):2575-2584. doi: 10.1212/WNL.0000000000003435. Epub 2016 Nov 9. PMID 27956565

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between July 2009 and May 2014 from 11 specialist NF1 academic clinics affiliated with the NF Clinical Trials Consortium.
Pre-assignment Details: After obtaining consent, participants were screened for study inclusion. If entry criteria were passed, they were randomized to study. All randomized participants were included in the primary efficacy analysis (baseline-to-post treatment) if they completed the baseline assessments.
Groups:
- Lovastatin: Oral lovastatin contained within in opaque capsules at a dose of 20mg a day (2 weeks) increased to a fixed dose of 40mg a day (14 weeks).
- Placebo: Look alike placebo pill with same dosing schedule as active lovastatin.
Period: Overall Study
Arm/Group | Lovastatin | Placebo
Started | 74 | 72
Completed | 67 | 56
Not Completed | 7 | 16
Not completed — Lost to Follow-up | 3 | 5
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Commenced contraindicated therapy | 0 | 2

BASELINE CHARACTERISTICS:
Population: Primary analyses of efficacy and safety were performed on the baseline to post-treatment data using the modified intention-to-treat population (defined as all subjects that had baseline data). Two participants from the placebo condition were excluded due to failure to complete baseline assessment.
Groups:
- Placebo: Look alike placebo capsule with same dosing schedule as active lovastatin.
- Total: Total of all reporting groups
Arm/Group | Lovastatin | Placebo | Total
Number analyzed (Participants) | 74 | 70 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74 | 70 | 144
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.5 (2.25) | 11.7 (1.95) | 11.6 (2.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 43 | 43 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 11 | 17
  White | 61 | 54 | 115
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 57 | 55 | 112
  Australia | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Paired Associate Learning (Cambridge Neuropsychological Test Automated Battery).
Description: A computerized test of visuospatial learning. Participants had to remember patterns associated with different locations on the screen, and during the test phase, as each pattern is presented, point to the appropriate location. The test starts at a very simple level and gradually increases in difficulty. Higher number of errors indicates poorer performance. Scale does not have a maximum range.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: Intention to treat using the modified intention-to-treat population (defined as all subjects that had baseline data). Missing post-treatment values were imputed using linear regression with age, sex and baseline values used as predictors (20 imputations).
Measure: Mean (Standard Error); unit: PAL Total Errors
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 73 | 68
PAL Total Errors
  Baseline | 15.8 (22.4) | 17.0 (15.4)
  Post-treatment | 10.3 (8.4) | 11.7 (11.7)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.51, ANCOVA

2. Primary Outcome: Score! (Test of Everyday Attention for Children)
Description: Score! is a measure of sustained attention. Participants were required to silently count a series of aurally presented tones and say the total number of tones counted at the end of each trial. The number of tones ranged from 9 to 15, with a total of 10 trials (range 0-10). Higher values represent better performance.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 73 | 66
Units on a scale
  Baseline | 6.0 (2.0) | 5.7 (2.4)
  Post-treatment | 7.3 (2.1) | 6.8 (2.5)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.33, ANCOVA

3. Secondary Outcome: Spatial Working Memory (Cambridge Neuropsychological Test Automated Battery)
Description: A computerized measure of spatial working memory. This task assessed the participant's ability to retain spatial information and to manipulate remembered items in working memory.
  In this test, participants were shown an array of boxes on a computer screen and they were required to search through the boxes for hidden tokens. One box at a time was touched until a blue token was found inside. Participants then commenced a new search for the next token. The key instruction was that, once a token had been located, that box would not be used again to hide another token.
  Unit of measure was between search errors, determined by the number of boxes a participant reopens in which a token had previously been found. Higher score indicated poorer performance. Scale does not have a maximum range.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 72 | 68
Errors
  Baseline | 47.0 (15.9) | 47.9 (16.2)
  Post-treatment | 40.4 (17.2) | 41.6 (17.0)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.86, ANCOVA

4. Secondary Outcome: Stockings of Cambridge (Cambridge Neuropsychological Test Automated Battery) Automated Battery).
Description: A computerized measure of spatial planning based on the "Tower of London" test. It required participants to move balls in a lower display to match a pattern shown in the upper display in a certain number of moves.
  More specifically, the participant was shown two displays containing three coloured balls. The displays were presented in such a way that they could be perceived as stacks of coloured balls held in socks suspended from a beam. The test administrator first demonstrated to the participant how to move the balls in the lower display to copy the pattern in the upper display and completed one demonstration problem, where the solution required one move. The participant then completed problems that increased in difficulty, from one through to five move problems.
  The unit of measure was the mean number of moves taken to complete a problem that could not be completed in less than five moves. The higher the score, the poorer the performance (range 5-12).
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Moves
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 71 | 66
Moves
  Baseline | 7.9 (1.4) | 8.0 (1.3)
  Post-treatment | 7.3 (1.4) | 7.9 (1.4)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.04, ANCOVA

5. Secondary Outcome: Stop Signal Task (Cambridge Neuropsychological Test Automated Battery)
Description: A computerized measure of inhibitory control. The participant quickly responded to an arrow stimulus by pressing one of two buttons (left or right), depending on the direction in which the arrow pointed on the screen. If an audio tone is present, the subject was supposed to withhold the response.
  The difficulty of the task was manipulated by altering the delay before a stop signal (auditory tone) was presented, known as the stop signal delay. The outcome from this measure was stop signal reaction time (last half of test), which was computed by subtracting the mean stop signal delay at which the participant was able to stop on 50% of trials from the mean reaction time on go trials. Poorer response inhibition was reflected by a larger stop signal reaction time. Scale does not have a maximum range.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 70 | 66
Milliseconds
  Baseline | 264.7 (98.7) | 237.2 (75.9)
  Post-treatment | 227.2 (87.2) | 227.0 (93.7)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.33, ANCOVA

6. Secondary Outcome: Sky Search (Test of Everyday Attention for Children)
Description: Sky Search is a measure of selective visual attention. Participants were presented with a A3 sheet with target stimuli (spaceships in identical pairs) randomly distributed among many distractors (spaceships in non-identical pairs). They were required to circle as many of the targets as possible as quickly as possible. The outcome measure (attention score), was a timing score reflecting the average time taken per target found. Higher scores represent poorer performance. Raw data are reported. Scale does not have a maximum range.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 74 | 66
Scores on a scale
  Baseline | 4.4 (1.7) | 5.0 (2.1)
  Post-treatment | 4.0 (2.0) | 4.4 (2.1)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.99, ANCOVA

7. Secondary Outcome: Sky Search DT (Test of Everyday Attention for Children)
Description: Sky Search DT is a test of divided attention. Children completed a parallel version of the Sky Search subtest while at the same time, silently counted the number of tones in a similar way to the Score! subtest. Higher scores represent poorer performance. Raw data are reported. Scale does not have a maximum range.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 73 | 66
Scores on a scale
  Baseline | 9.9 (15.5) | 9.6 (18.6)
  Post-treatment | 7.0 (15.6) | 6.6 (11.6)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.90, ANCOVA

8. Secondary Outcome: Creature Counting (Test of Everyday Attention for Children)
Description: Creature Counting is a measure of attentional control. Participants were required to count "creatures" from top of the page to the bottom, using arrows as cues to switch from counting up to counting down (and vice versa). There were seven testing trials. The outcome variable was the total number of correct trials (range 0-7). Higher scores represent better performances.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 74 | 66
Scores on a scale
  Baseline | 4.0 (2.2) | 3.8 (2.3)
  Post-treatment | 4.5 (1.9) | 4.6 (1.8)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.37, ANCOVA

9. Secondary Outcome: Commission Errors (Conners Continuous Performance Test, Second Edition; CPT-II)
Description: A computerised measure of impulse control. Letters were presented serially on a screen in a random order. All letters were considered target stimuli, except for the letter 'X' which is a non-target stimulus. Participants responded to target stimuli by pressing the space bar of a computer keyboard (90% of the stimuli) while withholding responses to non-target stimuli (10% of the test). Commission errors represented the number of times a participant incorrectly responded to the non-target (letter 'X'). T-scores are reported, as generated by the test software. Higher scores indicate poorer performances.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 74 | 64
T score
  Baseline | 57.5 (12.4) | 62.1 (17.2)
  Post-treatment | 58.8 (16.6) | 64.1 (18.4)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.49, ANCOVA

10. Secondary Outcome: Omission Errors (Conners Continuous Performance Test, Second Edition; CPT-II)
Description: A computerised measure of vigilance and concentration. Letters were presented serially on a screen in a random order. All letters were considered target stimuli, except for the letter 'X' which is a non-target stimulus. Participants responded to target stimuli by pressing the space bar of a computer keyboard (90% of the stimuli) while withholding responses to non-target stimuli (10% of the test). Omission errors represented the number of times a participant fails to respond to target letters (all other than 'X'). T-scores are reported, as generated by the test software. Higher scores indicate poorer performances.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 74 | 64
T score
  Baseline | 54.7 (10.5) | 56.9 (6.9)
  Post-treatment | 54.2 (10.5) | 55.5 (7.4)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.86, ANCOVA

11. Secondary Outcome: ADHD Inattentive Scale, Conners ADHD Scales
Description: Parent rated inattentive ADHD symptoms, based on Diagnostic and Statistical Manual of Mental Disorders criteria, 4th edition. T-scores are reported. Higher scores indicate increased ADHD-related symptoms. A score below 60 is considered healthy, 61-65 a possible significant problem, and 66+ is considered a significant problem.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 74 | 66
T score
  Baseline | 66.2 (12.6) | 64.0 (14.6)
  Post-treatment | 59.5 (13.2) | 61.1 (13.3)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.09, ANCOVA

12. Secondary Outcome: ADHD Hyperactive/Impulsive Scale, Conners ADHD Scales
Description: Parent rated hyperactive/impulsive ADHD symptoms, based on Diagnostic and Statistical Manual of Mental Disorders criteria, 4th edition.T-scores are reported. Higher scores indicate increased ADHD-related symptoms. A score below 60 is considered healthy, 61-65 a possible significant problem, and 66+ is considered a significant problem.
Time Frame: Baseline and Post-treatment (16 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 74 | 66
T score
  Baseline | 65.5 (14.2) | 62.9 (15.6)
  Post-treatment | 62.3 (15.4) | 62.3 (16.7)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.37, ANCOVA

13. Secondary Outcome: Controlled Oral Word Association Test
Description: A measure of verbal fluency. Participants were required to spontaneously produce as many words as they could, beginning with a designated letter in 60 seconds. Three letters were used. Higher scores represent better performances. Raw data are reported summing total words generated for all three letters. Scale does not have a maximum range.
Time Frame: Baseline and Post-treatment (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Total words
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 74 | 66
Total words
  Baseline | 22.2 (8.9) | 21.2 (8.6)
  Post-treatment | 22.2 (9.1) | 22.6 (8.9)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.18, ANCOVA

14. Secondary Outcome: Judgement of Line Orientation Test
Description: A test of visuospatial judgement. The test measured the participant's ability to match the angle and orientation of lines in space. There were 30 trial in total. Correct response in a trial was awarded one point (range 0-30). Higher scores represent better performances. Raw data are reported.
Time Frame: Baseline and Post-treatment (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Total correct responses
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 73 | 65
Total correct responses
  Baseline | 15.0 (6.6) | 14.6 (5.7)
  Post-treatment | 17.2 (7.0) | 16.7 (6.4)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.88, ANCOVA

15. Secondary Outcome: Behavior Rating Inventory of Executive Function Global Executive Composite
Description: A parent-rated questionnaire of executive behaviour assessing behavioral regulation (inhibit, shift, emotional control) and metacognition (initiate, working memory, plan/organize, organization of materials, self-monitoring). T-scores for the Global Executive Composite (overall summary score) are reported. Higher scores indicate poorer executive behaviors.
Time Frame: Baseline and Post-treatment (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 72 | 65
T score
  Baseline | 63.5 (11.5) | 61.4 (11.9)
  Post-treatment | 59.2 (13.2) | 58.8 (12.5)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.25, ANCOVA

16. Secondary Outcome: Object Assembly (WISC-III)
Description: A measure of visuoperceptual organization. Participants were required to rebuild an item puzzle based on disassembled pieces. Age scaled scores are reported, which have a population mean of 10 and standard deviation of 3 (range 1-19). Higher scores indicate better performances.
Time Frame: Baseline and Post-treatment (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 74 | 66
Scores on a scale
  Baseline | 6.6 (3.1) | 6.9 (3.0)
  Post-treatment | 7.8 (3.6) | 7.5 (3.3)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.20, ANCOVA

17. Secondary Outcome: Internalizing Behaviors, Behavior Assessment System for Children Second Edition
Description: A parent-reported questionnaire assessing internalizing behaviors of anxiety, depression and somatization. T-scores are reported. Higher scores indicate increased internalizing behaviors. A score below 60 is considered healthy, 61-65 a possible significant problem, and 66+ is considered a significant problem.
Time Frame: Baseline and Post-treatment (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 73 | 63
T score
  Baseline | 55.2 (12.6) | 53.8 (11.8)
  Post-treatment | 52.6 (12.6) | 52.5 (11.4)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.50, ANCOVA

18. Secondary Outcome: Internalizing Behaviors, Behavior Assessment System for Children Second Edition
Description: A self-reported questionnaire assessing internalizing behaviors such as anxiety and depression. T-scores are reported. Higher scores indicate increased internalizing behaviors. A score below 60 is considered healthy, 61-65 a possible significant problem, and 66+ is considered a significant problem.
Time Frame: Baseline and Post-treatment (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 73 | 63
T score
  Baseline | 50.9 (10.2) | 51.2 (8.7)
  Post-treatment | 47.9 (10.0) | 49.2 (8.5)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.33, ANCOVA

19. Secondary Outcome: Quality of Life Pediatric Quality of Life Inventory (PedsQL)
Description: Parent-rated questionnaire of psychosocial Quality of Life (including emotional, social and school functioning). Summary scores are reported. Higher scores indicate increased increased quality of life (range 0-100).
Time Frame: Baseline and Post-treatment (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 72 | 63
Scores on a scale
  Baseline | 62.8 (15.7) | 64.6 (18.1)
  Post-treatment | 69.2 (16.0) | 68.1 (16.6)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.30, ANCOVA

20. Secondary Outcome: Psychosocial Quality of Life PedsQL
Description: Self-rated questionnaire of psychosocial Quality of Life (including emotional, social and school functioning). Summary scores are reported. Higher scores indicate higher quality of life (range 0-100).
Time Frame: Baseline and Post-treatment (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 70 | 64
Scores on a scale
  Baseline | 67.2 (17.0) | 70.0 (18.1)
  Post-treatment | 62.6 (16.0) | 67.3 (17.0)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority; p = 0.73, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up assessment (24 weeks)
Description: Baseline to Follow-up assessment (24 weeks). Adverse events and serious adverse events were reported by organ system class.
Arm/Group | Lovastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/70
Serious Adverse Events (participants affected / at risk) | 6/74 | 1/70
Other Adverse Events (participants affected / at risk) | 65/74 | 59/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lovastatin (N=74) | Placebo (N=70)
Serious Adverse Event (General disorders) | 1 | 0
Serious Adverse Event (Blood and lymphatic system disorders) | 2 | 0
Serious Adverse Event (Hepatobiliary disorders) | 2 | 0
Serious Adverse Event (Musculoskeletal and connective tissue disorders) | 1 | 0
Serious Adverse Event (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lovastatin (N=74) | Placebo (N=70)
General (General disorders) | 29 | 23
Cardiovascular (Cardiac disorders) | 7 | 7
Gastrointestinal (Gastrointestinal disorders) | 33 | 32
Hematologic (Blood and lymphatic system disorders) | 10 | 12
Hepatobiliary (Hepatobiliary disorders) | 3 | 4
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 21 | 17
Nervous (Nervous system disorders) | 19 | 26
Respiratory (Respiratory, thoracic and mediastinal disorders) | 32 | 26
Skin/appendages (Skin and subcutaneous tissue disorders) | 21 | 14
Special senses - Eye (Eye disorders) | 6 | 3
Special Senses - Ear (Ear and labyrinth disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2011-05-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT00853580/Prot_000.pdf
  • Statistical Analysis Plan (2011-05-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT00853580/SAP_001.pdf
  • Informed Consent Form (2013-01-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT00853580/ICF_002.pdf